CLINICAL TRIAL: NCT05388968
Title: Pathogen Detection by Metatranscriptomic Next Generation Sequencing in the Trophoblast Collected in Women Carrying a Fetus With Increasing Nuchal Translucency in the First Trimester of Pregnancy
Brief Title: Metatranscriptomic Next Generation Sequencing in First Trimester Trophoblast With Increased Fetal Nuchal Translucency (METAHCN)
Acronym: METAHCN
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Pathogen Discovery Laboratory (Unknown); Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: APHP211328
Record Dates: First submitted 2022-05-02; First posted 2022-05-24 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Increased Nuchal Translucency in the First Trimester of Pregnancy
Keywords: nuchal translucency; metatranscriptomic; next generation sequencing; metagenomic; trophoblast; high throughput sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Nuchal translucency with no genetic abnormalities: Pregnant women between 11 and 14 weeks with a fetus showing a nuchal translucency > 3.5 mm and no genetic abnormalities with array CGH.
  Interventions: Biological: Metatranscriptomic; Diagnostic Test: Specific microbiologic diagnosis
- Nuchal translucency with genetic abnormalities: Pregnant women between 11 and 14 weeks with a fetus showing a nuchal translucency > 3.5 mm and a genetic abnormalities at array CGH.
  Interventions: Biological: Metatranscriptomic; Diagnostic Test: Specific microbiologic diagnosis
- Genetic abnormalities: Pregnant women between 11 and 14 weeks with a fetus showing a nuchal translucency < 3.5 mm and a suspicion of genetic abnormalities
  Interventions: Biological: Metatranscriptomic; Diagnostic Test: Specific microbiologic diagnosis

INTERVENTIONS:
Biological: Metatranscriptomic — Analysis with metatranscriptomic next generation sequencing of trophoblast obtained by chorionic villi sampling
Diagnostic Test: Specific microbiologic diagnosis — If a microorganism is detected by metatranscriptomic NGS, specific diagnosis (PCR and serology) will be done in maternal and neonatal samples (blood, urine, saliva)

SUMMARY:
The study is based on the hypothesis that increased nuchal translucency may be associated with a materno fetal infection and that the pathogen responsible for this infection could be identify with metatranscriptomic next-generation sequencing in the trophoblast tissue.

DETAILED DESCRIPTION:
Nuchal translucency > 3.5 mm in the first trimester of pregnancy is due to fluid accumulation in the subcutaneous tissue in the nuchal area. This is seen in around 1% of all pregnancies. Increased nuchal translucency is explained by a chromosomic abnormality (mainly Down syndrome) in 30 to 40% of cases. Therefore, the state of the art is to perform an array CGH on chorionic villi sampling. Cases of nuchal translucency that are not explained by a chromosomic abnormality may be associated: with fetal defect (heart, congenital diaphragmatic hernia) in 10% of cases, with genetic disease in 4% of cases or with miscarriage or fetal death of unknown etiology in 18% of cases.

The etiology of increased nuchal translucency remains unknown in more than 50% of the cases. It could be linked to inflammation or reflect an infection but this latter association has been rarely studied. This association was suggested in a study reporting serology of CMV, toxoplasmosis or B19 parvovirus primary infections in pregnant women carrying a fetus with increased nuchal translucency. In those rare cases, the microorganism was not searched directly in the trophoblast tissue. In the investigators' center, the investigators describe in a context of maternal primary infection, one case of increased nuchal translucency with a positive CMV PCR in the trophoblast tissue collected at 12 weeks. Other pathogens yet not identified might be associated with increased nuchal translucency.

Metatranscriptomic next generation sequencing (mNGS) allows to search for any pathogens without a priori. It is therefore a powerful technic to study this potential association between increased nuchal translucency and infection.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Singleton pregnancy
* First trimester (11 GA+0D to 13 GA+6D)
* Carrying a fetus with a nuchal translucency > 3.5 mm for which a chorionic villi sampling is performed OR a suspicion of genetic abnormalities for which a chorionic villi sampling is performed
* Delivery planned at Necker hospital
* Not opposed to participation

Exclusion Criteria

* Age <18 years
* no health insurance
* difficulties in understanding the French language
* chronic infection (HIV, HBV, HVC and HTLV-1)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women consulting in the prenatal diagnosis Unit of the University Hospital Necker-Enfants-malades
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
microorganisms (viruses, bacteria, or parasites) in trophoblast samples | At inclusion, 11-14 weeks of pregnancy
  Identification by metatranscriptomic NGS, from women carrying a fetus with nuchal translucency (group 1) and in controls (group 2 and 3)

SECONDARY OUTCOMES:
Miscarriage | at termination of pregnancy (assessed up to 7 months)
  Comparison in group 1 of the proportion of miscarriageaccording to the presence or not of a microorganism in the trophoblast.
intrauterine death | at termination of pregnancy (assessed up to 7 months)
  Comparison in group 1 of the proportion of intrauterine death according to the presence or not of a microorganism in the trophoblast.
fetal abnormalities | at delivery
  Comparison in group 1 of the proportion of fetal abnormalities, according to the presence or not of a microorganism in the trophoblast.
Gestational age | at delivery
  Comparison in group 1 of gestational age at birth, according to the presence or not of a microorganism in the trophoblast.
birth weight | at delivery
  Comparison in group 1 of birth weight, according to the presence or not of a microorganism in the trophoblast.
Detection of the microorganism identified by metatranscriptomic NGS by conventional diagnostic method in maternal samples | at inclusion
  Amplification by real time PCR of the microorganism identified by metatranscriptomic NGS in maternal blood, urine, saliva and amniotic fluid if available
Detection of the microorganism identified by metatranscriptomic NGS by conventional diagnostic method in maternal samples | at inclusion
  specific serology to identify a maternal primary infection with the microorganism detected by metatranscriptomic NGS
Detection of the microorganism identified by metatranscriptomic NGS by conventional diagnostic method in neonatal samples | 3 days after birth
  Amplification by real time PCR of the microorganism identified by metatranscriptomic NGS in neonatal blood, urine, saliva
Detection of the microorganism identified by metatranscriptomic NGS by conventional diagnostic method in neonatal samples | 3 days after birth
  specific serology to identify a maternal primary infection with the microorganism detected by metatranscriptomic NGS

CONTACTS AND LOCATIONS:
Overall Officials: Marianne LERUEZ-VILLE, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Yves Ville, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Necker - Enfants malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sebire NJ, Bianco D, Snijders RJ, Zuckerman M, Nicolaides KH. Increased fetal nuchal translucency thickness at 10-14 weeks: is screening for maternal-fetal infection necessary? Br J Obstet Gynaecol. 1997 Feb;104(2):212-5. doi: 10.1111/j.1471-0528.1997.tb11047.x. PMID 9070141
- [Background] Faure-Bardon V, Fourgeaud J, Guilleminot T, Magny JF, Salomon LJ, Bernard JP, Leruez-Ville M, Ville Y. First-trimester diagnosis of congenital cytomegalovirus infection after maternal primary infection in early pregnancy: feasibility study of viral genome amplification by PCR on chorionic villi obtained by CVS. Ultrasound Obstet Gynecol. 2021 Apr;57(4):568-572. doi: 10.1002/uog.23608. Epub 2021 Mar 9. PMID 33533526
- [Background] Regnault B, Bigot T, Ma L, Perot P, Temmam S, Eloit M. Deep Impact of Random Amplification and Library Construction Methods on Viral Metagenomics Results. Viruses. 2021 Feb 7;13(2):253. doi: 10.3390/v13020253. PMID 33562285
- [Background] Bilardo CM, Timmerman E, Pajkrt E, van Maarle M. Increased nuchal translucency in euploid fetuses--what should we be telling the parents? Prenat Diagn. 2010 Feb;30(2):93-102. doi: 10.1002/pd.2396. PMID 20077440